CLINICAL TRIAL: NCT06104644
Title: Deucravacitinib in Routine Clinical Practice: A 5-year, Multicenter, Prospective, Non-Interventional Cohort Study to Evaluate Effectiveness and Quality of Life in Patients With Moderate-to-Severe Plaque Psoriasis in Germany (DELPHIN)
Brief Title: A Study to Evaluate Deucravacitinib in Participants With Moderate-to-Severe Plaque Psoriasis in Germany
Acronym: DELPHIN
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM011-250
Record Dates: First submitted 2023-10-06; First posted 2023-10-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — deucravacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Moderate-to-severe plaque psoriasis
  Interventions: Drug: Deucravacitinib

INTERVENTIONS:
Drug: Deucravacitinib — Non-interventional observational study of patients receiving treatment with commercially available deucravacitinib 6 mg once daily according to the Summary of Product Characteristics

SUMMARY:
The purpose of this observational study is to describe the effectiveness of deucravacitinib treatment and quality of life in adults with moderate-to-severe plaque psoriasis in routine clinical practice in Germany over a 5-year period

ELIGIBILITY:
Inclusion Criteria:

* Patients with a physician-reported diagnosis of moderate-to-severe plaque psoriasis initiating deucravacitinib according to approved label in the European Union
* The decision upon treatment with deucravacitinib must have been made before enrollment and independently of this non-interventional observational study
* Patient is at least 18 years of age at the time of treatment decision
* Patient provided written informed consent to participate in the study

Exclusion Criteria:

* Any contraindications according to the approved deucravacitinib Summary of Product Characteristics
* Prior treatment with deucravacitinib
* Simultaneous participation in an interventional clinical trial for moderate-to-severe psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with moderate-to-severe plaque psoriasis in Germany
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving an absolute Psoriasis Area Severity Index (aPASI) score ≤ 3 at Week 24 or nearest visit | Approximately 24 weeks after treatment initiation (data to be collected at visit nearest to this timepoint)

SECONDARY OUTCOMES:
Effectiveness of deucravacitinib treatment measured by the number of participants who achieve an absolute Psoriasis Area Severity Index (aPASI) score ≤ 3 and ≤ 6 | 5 years
Effectiveness of deucravacitinib treatment measured by the number of participants who achieve Psoriasis Area Severity Index (PASI) 75/90/100 | 5 years
Effectiveness of deucravacitinib treatment measured by the number of participants who achieved static Physician's Global Assessment (sPGA) 0/1 and change in sPGA over time | 5 years
Effectiveness of deucravacitinib treatment measured by body surface area (BSA) affected by psoriasis and changes in BSA from baseline and over time | 5 years
Effectiveness of deucravacitinib treatment in sensitive body areas measured by Physician's Global Assessment (PGA) for the genital area | 5 years
Effectiveness of deucravacitinib treatment in sensitive body areas measured by Physician's Global Assessment (PGA) for the intertriginous areas | 5 years
  Including but not limited to axilla, popliteal fossa, inguinal, genital, submammary, anal region
Effectiveness of deucravacitinib treatment in sensitive body areas measured by palmoplantar psoriasis Physician's Global Assessment (pp-PGA) for the palmoplantar area | 5 years
Effectiveness of deucravacitinib treatment in sensitive body areas measured by target Nail Psoriasis Severity Index (NAPSI) for the nails | 5 years
Effectiveness of deucravacitinib treatment in sensitive body areas measured by scalp-specific Physician's Global Assessment (ss-PGA) for the scalp | 5 years
Treatment modalities and patient's satisfaction with deucravacitinib therapy measured by the Treatment Satisfaction Questionnaire for Medication (TSQM)-9 | 5 years
Treatment modalities and patient's satisfaction with deucravacitinib therapy measured by the persistence of deucravacitinib therapy | 5 years
  Time from therapy initiation until discontinuation visualized using Kaplan-Meier methods
Treatment modalities and patient's satisfaction with deucravacitinib therapy measured by reasons for therapy discontinuation | 5 years
  Discontinuation of deucravacitinib defined as a treatment interruption of >90 days with or without resumption of deucravacitinib treatment, with or without start of a follow-up therapy
Patient-reported outcomes measured by the Dermatology Life Quality Index (DLQI) | 5 years
Patient-reported outcomes evaluating pruritus measured by the Itch Numeric Rating Scale (NRS) | 5 years
Patient-reported outcomes measured by the Patient Benefit Index standard version (PBI-S) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Germany (2):
  - Dermatologische Spezial- und Schwerpunktpraxis Selters, Selters, Rhineland-Palatinate
  - Local Institution - 0001, Selters

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts